CLINICAL TRIAL: NCT02600403
Title: Reversible Structural and Functional Changes After Intraocular Pressure Reduction in Patients With Glaucoma
Brief Title: Are There Changes in the Nerve Fiber Layer (NFL) After Lowering of Eye Pressure?
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, George L. Spaeth MD, MD, Wills Eye
Other Study IDs: 11-058
Record Dates: First submitted 2015-08-10; First posted 2015-11-09 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Glaucoma
Keywords: Visual Evoked Potentials; Optical Coherence Tomography; Visual Fields
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence; Evoked Potentials, Visual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- IOP between 22-32 mmHg: Forty four (44) patients with intraocular pressure between 22 and 32 millimeters (mmHg) of mercury will undergo Optical Coherence Tomography (OCT); Visual Evoked Potential (VEP); and Humphrey Visual Field (HVF).
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT); Diagnostic Test: Visual evoked potential (VEP); Diagnostic Test: Humphrey Visual Field (HVF)
- IOP greater than 32 mmHg: Six (6) patients with intraocular pressure greater than 32 millimeters of mercury (mmHg) will undergo Optical Coherence Tomography (OCT); Visual Evoked Potential (VEP); and Humphrey Visual Field (HVF).
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT); Diagnostic Test: Visual evoked potential (VEP); Diagnostic Test: Humphrey Visual Field (HVF)
- IOP less than 22 mmHg: Eleven (11) patients with stable intraocular pressure (less than 22 millimeters of mercury (mmHg)) on ophthalmic solutions (eye drops) will undergo Optical Coherence Tomography (OCT); Visual Evoked Potential (VEP); and Humphrey Visual Field (HVF).
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT); Diagnostic Test: Visual evoked potential (VEP); Diagnostic Test: Humphrey Visual Field (HVF)

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography (OCT) — Optical Coherence Tomography (OCT) is a machine that scans eyes and has the capability of measuring thickness of various layers of the retina and nerve fiber layer (NFL).
  Other Names: OCT
Diagnostic Test: Visual evoked potential (VEP) — Visual Evoked Potential (VEP) is an imaging system that measures electrical activity from the eye to the brain by using electrodes placed on forehead and back of the head similar to electroencephalogram (EEG).
  Other Names: VEP
Diagnostic Test: Humphrey Visual Field (HVF) — Humphrey Visual Field (HVF) is a test done to evaluate how much peripheral (side) vision has been lost due to glaucoma.
  Other Names: VF

SUMMARY:
The aim of this study was to evaluate structural and functional improvement after lowering intraocular pressure (IOP) in patients with glaucoma using Spectral Domain Optical Coherence Tomography (SD-OCT), Visual Field (VF) testing, and Visual Evoked Potential (VEP).

DETAILED DESCRIPTION:
Glaucoma exhibits characteristic changes to the optic nerve in the back of the eye. The optic nerve is formed when fibers that overlay the retina come together. This layer is called the retinal nerve fiber layer (RNFL).

Optical Coherence Tomography (OCT) is a machine that scans eyes and has the capability of measuring thickness of various layers in the retina and RNFL. This provides important anatomical information.

VEP (visual evoked potential) is an imaging system that measures electrical signals from the eye to the brain by using electrodes placed on the forehead and back of head. This is similar in principal to an electrocardiogram of the heart.

Visual field testing is done to evaluate the extent of side vision loss caused by various diseases of the eye, including glaucoma. This testing is performed as you stare at a small light directly in front of your eye while lights flash one at a time in every direction on a screen surrounding the central light. You push a button each time you see a flash out of the corner of your eye.

Lowering intraocular pressure (IOP) in the eye has been shown to result in reversal of glaucoma changes of the optic nerve in some patients. It has also been suggested that improvement in function (visual field) has been associated with improved optic nerve appearance.

This study seeks to provide evidence for reversal of disc appearance and visual function following IOP lowering interventions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with glaucoma (primary open-angle glaucoma, angle recession glaucoma, exfoliation syndrome glaucoma, pigmentary glaucoma and chronic angle closure glaucoma) in whom a pressure-lowering intervention was conducted

Exclusion Criteria:

* Inability to obtain reliable field or optical coherence tomography pre-intervention
* Visual acuity less than 20/40,
* Age <18 or >90 years,
* Other cause for visual field loss not glaucoma, that is, visual field loss due to cataract optic neuropathies, retinal disease
* Spherical equivalent refractive error > +5.00 Diopters and > 3.00 Diopters cylinder
* Concomitant cataract and glaucoma surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients with intraocular pressure (IOP) between 22 and 32 millimeters of mercury (mm HG); greater than 32 mm HG; and with stable IOPs (control group).
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Spaeth, MD, Principal Investigator — Wills Eye

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jindal AP, Fleischman D, Leiby B, Spaeth GL, Myers JS, Katz LJ. Effects of acutely lowering intraocular pressure on the results of multifocal visual evoked potential testing. Acta Ophthalmol. 2011 Nov;89(7):e550-4. doi: 10.1111/j.1755-3768.2011.02177.x. Epub 2011 May 23. PMID 21599873
- [Background] Waisbourd M, Ahmed OM, Molineaux J, Gonzalez A, Spaeth GL, Katz LJ. Reversible structural and functional changes after intraocular pressure reduction in patients with glaucoma. Graefes Arch Clin Exp Ophthalmol. 2016 Jun;254(6):1159-66. doi: 10.1007/s00417-016-3321-2. Epub 2016 Mar 19. PMID 26995555

RESULTS

PARTICIPANT FLOW:
Groups:
- Glaucoma Subjects With IOP 22-32 mmHg: Forty four (44) patients will have testing done using optical coherence tomography (OCT), visual evoked potential (VEP) and visual field (VF).
  Testing will be repeated at 1-2 months, 4-6 months and 9-12 months after the initial eye pressure intervention (follow-up testing will be one (1) visual field test, two (2) OCT's and one (1) VEP).
  Optical Coherence Tomography (OCT): Optical Coherence Tomography (OCT) is a machine that scans the eyes and has the capability of measuring the thickness of the various layers of the retina and NFL.
  Visual Evoked Potential (VEP): Visual Evoked Potential (VEP) is an imaging system that measures the electrical signal from the eye to the brain by using electrodes placed on the forehead and back of the head.
  Visual Field: Visual field testing is done to evaluate the extent of side vision loss a patient has with various diseases of the eye, including glaucoma.
- Glaucoma Subjects With IOP >32 mmHg: Six (6) patients will have testing done using optical coherence tomography (OCT), Visual Evoked Potential (VEP) and visual field (VF).
  This testing will be repeated one (1) hour, one (1) day and three (3) months following the eye pressure lowering intervention.
  Optical Coherence Tomography (OCT): Optical Coherence Tomography (OCT) is a machine that scans the eyes and has the capability of measuring the thickness of the various layers of the retina and NFL.
  Visual Evoked Potential (VEP): Visual Evoked Potential (VEP) is an imaging system that measures the electrical signal from the eye to the brain by using electrodes placed on the forehead and back of the head.
  Visual Field: Visual field testing is done to evaluate the extent of side vision loss a patient has with various diseases of the eye, including glaucoma.
- Control Glaucoma Subjects: Eleven (11) patients will have testing done using optical coherence tomography (OCT), Visual Evoked Potential (VEP) and visual field (VF).
  Testing will be repeated at 1-2 months, 4-6 months and 9-12 months after the initial testing was completed.
  Optical Coherence Tomography (OCT): Optical Coherence Tomography (OCT) is a machine that scans the eyes and has the capability of measuring the thickness of the various layers of the retina and NFL.
  Visual Evoked Potential (VEP): Visual Evoked Potential (VEP) is an imaging system that measures the electrical signal from the eye to the brain by using electrodes placed on the forehead and back of the head.
  Visual Field: Visual field testing is done to evaluate the extent of side vision loss a patient has with various diseases of the eye, including glaucoma.
Period: Overall Study
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Started | 44 | 6 | 11
Completed | 44 | 6 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Glaucoma Subjects With Intra-ocular Pressure 22-32 mmHg: Forty four (44) patients will have testing done using optical coherence tomography (OCT), visual evoked potential (VEP) and visual field (VF).
  Testing will be repeated at 1-2 months, 4-6 months and 9-12 months after the initial eye pressure intervention (follow-up testing will be one (1) visual field test, two (2) OCT's and one (1) VEP).
  Optical Coherence Tomography (OCT): Optical Coherence Tomography (OCT) is a machine that scans the eyes and has the capability of measuring the thickness of the various layers of the retina and NFL.
  Visual Evoked Potential (VEP): Visual Evoked Potential (VEP) is an imaging system that measures the electrical signal from the eye to the brain by using electrodes placed on the forehead and back of the head.
  Visual Field: Visual field testing is done to evaluate the extent of side vision loss a patient has with various diseases of the eye, including glaucoma.
- Glaucoma Subjects With Intra-ocular Pressure >32 mmHg: Six (6) patients will have testing done using optical coherence tomography (OCT), Visual Evoked Potential (VEP) and visual field (VF).
  This testing will be repeated one (1) hour, one (1) day and three (3) months following the eye pressure lowering intervention.
  Optical Coherence Tomography (OCT): Optical Coherence Tomography (OCT) is a machine that scans the eyes and has the capability of measuring the thickness of the various layers of the retina and NFL.
  Visual Evoked Potential (VEP): Visual Evoked Potential (VEP) is an imaging system that measures the electrical signal from the eye to the brain by using electrodes placed on the forehead and back of the head.
  Visual Field: Visual field testing is done to evaluate the extent of side vision loss a patient has with various diseases of the eye, including glaucoma.
- Total: Total of all reporting groups
Arm/Group | Glaucoma Subjects With Intra-ocular Pressure 22-32 mmHg | Glaucoma Subjects With Intra-ocular Pressure >32 mmHg | Control Glaucoma Subjects | Total
Number analyzed (Participants) | 44 | 6 | 11 | 61
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [27 to 84] | 65.5 [55 to 75] | 60 [45 to 79] | 64.5 [27 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 1 | 3 | 23
  Male | 25 | 5 | 8 | 38

OUTCOME MEASURES:

1. Primary Outcome: Visual Field Mean Deviation
Description: Visual field mean deviation as measured in decibels (dB) is the amount of visual field loss compared to age matched controls (people with no eye diseases or visual field loss). Brightness of the flashes of light used to test peripheral vision during a visual field test is measured in decibels. Brighter light has lower number in decibels. The dimmer the light, the higher the number in decibels with a range of 0 to 40 dB.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: dB (decibels)
Groups:
- Glaucoma Subjects With IOP 22-32 mmHg: Forty four (44) patients will have optical coherence tomography (OCT), visual evoked potential (VEP) and visual field (VF) repeated at 1-2 months, 4-6 months and 9-12 months after initial eye pressure intervention (follow-up testing will be one (1) visual field test, two (2) OCT's and one (1) VEP).
  Optical Coherence Tomography (OCT): is a series of eye scans with capability of measuring thickness of the various layers of the retina and RNFL.
  Visual Evoked Potential (VEP): is a system that measures electrical signals from the eye to the brain by electrodes placed on the forehead and back of the head.
  Visual Field: testing is done to evaluate extent of side vision loss from various diseases of the eye, including glaucoma.
- Glaucoma Subjects With IOP >32 mmHg: Six (6) patients will have optical coherence tomography (OCT), visual evoked potential (VEP) and visual field (VF) repeated at 1-2 months, 4-6 months and 9-12 months after initial eye pressure intervention (follow-up testing will be one (1) visual field test, two (2) OCT's and one (1) VEP).
  Optical Coherence Tomography (OCT): is a series of eye scans with capability of measuring thickness of the various layers of the retina and RNFL.
  Visual Evoked Potential (VEP): is a system that measures electrical signals from the eye to the brain by electrodes placed on the forehead and back of the head.
  Visual Field: testing is done to evaluate extent of side vision loss from various diseases of the eye, including glaucoma.
- Control Glaucoma Subjects: Eleven (11) patients will have optical coherence tomography (OCT), visual evoked potential (VEP) and visual field (VF) repeated at 1-2 months, 4-6 months and 9-12 months after initial eye pressure intervention (follow-up testing will be one (1) visual field test, two (2) OCT's and one (1) VEP).
  Optical Coherence Tomography (OCT): is a series of eye scans with capability of measuring thickness of the various layers of the retina and RNFL.
  Visual Evoked Potential (VEP): is a system that measures electrical signals from the eye to the brain by electrodes placed on the forehead and back of the head.
  Visual Field: testing is done to evaluate extent of side vision loss from various diseases of the eye, including glaucoma.
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Number analyzed (Participants) | 44 | 6 | 11
dB (decibels)
  Pre-operative | -8.7 (8.2) | -13.3 (9.7) | -13.2 (10.6)
  Follow up 1 | -8.3 (7.84) | -14.1 (10.15) | -8.6 (7.87)
  Follow up 2 | -8.5 (7.19) | -13.8 (10.66) | -9.4 (7.68)
  Follow up 3 | -9.4 (8.5) | -14.8 (12.2) | -10.4 (7.4)

2. Primary Outcome: Retinal Nerve Fiber Layer (RNFL) Thickness Measurement
Description: Retinal nerve fiber layer (RNFL) thickness in different quadrants of optic nerve and macula are measured pre and postoperatively to evaluate structural changes.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Number analyzed (Participants) | 44 | 6 | 11
um
  Pre-operative | 75.5 (16.1) | 74.3 (10.2) | 70.4 (11.7)
  Follow up 1 | 74.9 (15.22) | 76 (9.08) | 69.4 (2.05)
  Follow up 2 | 73.8 (20.53) | 75.2 (9.75) | 68.9 (0)
  Follow up 3 | 74.7 (11.03) | 74.1 (10.68) | 67.4 (0.5)

3. Primary Outcome: Average Cup to Disc Ratio
Description: Cup to disc ratio is used to evaluate structural changes comparing the size of the cup to the size of the disc during dilated ophthalmic examination. High eye pressure can cause the cup to enlarge, closer to the size of the disc. This measurement is used to follow progression in glaucoma. A normal range for cup to disc ratio would be 0.0 to 0.4. Advanced glaucoma would be 0.8 to 0.9 cup to disc ratio.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Number analyzed (Participants) | 44 | 6 | 11
ratio
  Pre-operative | 0.71 (0.12) | 0.76 (0.17) | 0.76 (0.09)
  Follow up 1 | 0.69 (0.17) | 0.74 (0.20) | 0.77 (0.034)
  Follow up 2 | 0.68 (0.20) | 0.72 (0.19) | 0.75 (0)
  Follow up 3 | 0.68 (0.08) | 0.72 (0.22) | 0.77 (0.01)

4. Primary Outcome: Visual Evoked Potential Amplitudes
Description: VEP amplitudes at high contrast as measured in microvolts (μV). Electroencephalogram (EEG) measures electrical activity in the brain. VEP measures electrical activity in areas of the brain responsible for vision by using EEG electrodes. The amplitude measurement is the peak of the energy generated (strongest strength of the signal) from the eye's response to the visual stimulus during the VEP.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: micro volts (uV)
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Number analyzed (Participants) | 44 | 6 | 11
micro volts (uV)
  Pre-operative Amplitude High Contrast | 12.7 (14.4) | 10.7 (5.4) | 12.1 (8.33)
  Follow up 1 Amplitude High Contrast | 12.1 (6.73) | 9.5 (1.78) | 12.5 (8.6)
  Follow up 2 Amplitude High Contrast | 12.4 (3.34) | 9.2 (4.56) | NA (NA) — values not calculated for visits 2 and 3 due to missing data. patients in this group did not return for all follow-up visits.
  Follow up 3 Amplitude High Contrast | 11.8 (4.3) | 12.1 (5.5) | NA (NA) — values not calculated for visits 2 and 3 due to missing data

5. Primary Outcome: Visual Evoked Potential Latency
Description: VEP latency at high contrast as measured in milliseconds (ms). Electroencephalogram (EEG) measures electrical activity in the brain. VEP measures electrical activity in areas of the brain responsible for vision by using EEG electrodes. VEP latencies measure the duration in time of the energy generated (duration of the signal) from the eye's response to a visual stimulus during the VEP.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Milli-seconds (ms)
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Number analyzed (Participants) | 44 | 6 | 11
Milli-seconds (ms)
  Pre-operative | 126.1 (14.67) | 117.0 (20.25) | 114.1 (19.70)
  Follow up 1 Latency High Contrast | 110.1 (18.56) | 125.7 (3.40) | 139.8 (1.95)
  Follow up 2 Latency High Contrast | 123.1 (19.95) | 124.2 (13.36) | NA (NA) — values not calculated for visits 2 and 3 due to missing data
  Follow up 3 Latency High Contrast | 118.8 (3.23) | 127.5 (13.76) | NA (NA) — values not calculated for visits 2 and 3 due to missing data

6. Primary Outcome: Visual Field
Description: Visual field pattern standard deviation in decibels (dB). Visual field results compare visual field loss to age matched controls (people with no eye diseases or visual field loss). Brightness of the flashes of light used to test peripheral vision during a visual field test is measured in decibels. With a localized defect in the visual field, pattern standard deviation (PSD) quantifies amount of loss and progression of glaucoma when in the beginning stages of the disease.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
Number analyzed (Participants) | 44 | 6 | 11
dB
  Pre-operative | 4.9 (3.57) | 6.3 (3.33) | 6.8 (3.99)
  Follow up 1 | 5.0 (3.54) | 4.0 (2.95) | 5.8 (4.42)
  Follow up 2 | 5.1 (3.63) | 5.0 (2.97) | 6.7 (4.80)
  Follow up 3 | 5.0 (4.00) | 4.1 (2.25) | 6.4 (5.04)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Study imaging and tests (visual field, optical coherence tomography, visually evoked potentials) involved non-invasive techniques. Results were compared between visits. No adverse event data was captured or reported.
Arm/Group | Glaucoma Subjects With IOP 22-32 mmHg | Glaucoma Subjects With IOP >32 mmHg | Control Glaucoma Subjects
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 0/44 | 0/6 | 0/11

LIMITATIONS AND CAVEATS:
Small sample size. Patients grouped by baseline intraocular pressure not by intervention. Inconsistent follow-up times. Subset of moderate to advanced glaucoma precluding possibility of reversible VEP changes in earlier stages of glaucoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No